CLINICAL TRIAL: NCT00415376
Title: A Pilot Study of the Efficacy of Levetiracetam in Patients With Seizures From Brain Metastases
Brief Title: Levetiracetam in Treating Patients With Seizures Caused by Brain Metastases
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to accrue subjects
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: CDR0000520380; NU-05CC11; NU-1398-032; UCB-NU-05CC11
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Brain and Central Nervous System Tumors; Seizure; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: seizure; adult tumors metastatic to brain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Central Nervous System Neoplasms; Seizures; Brain Neoplasms | interventions — Levetiracetam

INTERVENTIONS:
Drug: levetiracetam
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Anticonvulsant drugs, such as levetiracetam, may help control seizures caused by brain metastases.

PURPOSE: This clinical trial is studying the side effects and how well levetiracetam works in treating patients with seizures caused by brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the optimal dose of levetiracetam required to control seizures from brain metastases in patients with solid tumors.
* Determine the frequency of side effects and tolerability of this drug when used to control seizures in these patients.
* Determine any improvement in antiepileptic drug-associated symptoms in these patients.

OUTLINE: This is a pilot study. Patients are stratified according to baseline seizures (yes vs no) and/or baseline antiepileptic drugs (AEDs) (yes vs no). Patients are assigned to 1 of 3 treatment groups.

* Group I (patients with no active baseline seizures): Patients receive oral levetiracetam twice daily beginning on day 1.
* Group II (patients requiring IV AEDs for baseline seizure control): Patients receive oral levetiracetam (instead of their current anticonvulsant therapy) twice daily beginning on day 1, after their presenting condition has stabilized.
* Group III (patients with active seizures controlled by other concurrent anticonvulsant monotherapy): Patients receive oral levetiracetam (instead of their current anticonvulsant therapy) twice daily beginning on day 1. Treatment with the other anticonvulsant drug is tapered beginning on day 3 as directed by the treating physician.

In all groups, treatment continues for up to 6 months in the absence of uncontrolled seizures or unacceptable toxicities.

During study therapy, patients maintain a seizure log that tracks frequency and type of seizures. Any patient who experiences a breakthrough seizure or multiple auras receives increasing doses of oral levetiracetam until the maximum dose is reached. Patients who continue to have seizures at the maximum dose level receive a second antiseizure medication at the discretion of the treating physician.

Quality of life is assessed by the Fundamental Assessment of Cancer Treatment-Brain questionnaire at baseline and at 2 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Pathological confirmation of brain metastasis is not required provided the clinical and neuroradiographic picture is typical
* Has had at least one prior seizure due to brain metastasis

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 12 weeks
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* BUN < 5 times upper limit of normal (ULN)
* Creatinine < 5 times ULN
* Bilirubin < 1.5 times ULN
* AST and ALT ≤ 3 times ULN
* Alkaline phosphatase ≤ 2 times ULN
* No allergy to levetiracetam

PRIOR CONCURRENT THERAPY:

* Prior levetiracetam allowed provided it was initiated within the past 14 days
* Other concurrent anticonvulsant monotherapy allowed provided therapy was initiated within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07

PRIMARY OUTCOMES:
Seizure control (lack of seizure activity)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Raizer, MD, Principal Investigator — Robert H. Lurie Cancer Center